CLINICAL TRIAL: NCT07182097
Title: Effects of Intraoperative Fentanyl vs. Remifentanil on Postoperative Bowel Function and Pain Outcomes in Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Fentanyl vs. Remifentanil in Laparoscopic Cholecystectomy: Effects on Bowel Function and Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, MUSTAFA BÜYÜKCAVLAK, Specialist in Anesthesiology and Intensive Care, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 364/2025
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Bowel Function; Postoperative Pain
Keywords: postoperative pain; postoperative ileus; postoperative bowel function; fentanyl; remifentanil
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl Group (Active Comparator): Patients will receive fentanyl 2 µg/kg IV bolus at induction, followed by a continuous infusion of 1-2 µg/kg/h during maintenance of anesthesia. Standard anesthesia will be provided with propofol, rocuronium, and sevoflurane.
  Interventions: Drug: Fentanyl 2 µg/kg IV bolus + 1-2 µg/kg/h infusion during anesthesia
- Remifentanil Group (Active Comparator): Patients will receive remifentanil 1 µg/kg IV bolus at induction, followed by a continuous infusion of 0.1-1 µg/kg/min during maintenance of anesthesia. Standard anesthesia will be provided with propofol, rocuronium, and sevoflurane.
  Interventions: Drug: Remifentanil 1 µg/kg IV bolus + 0.1-1 µg/kg/min infusion during anesthesia

INTERVENTIONS:
Drug: Fentanyl 2 µg/kg IV bolus + 1-2 µg/kg/h infusion during anesthesia — Patients will receive fentanyl 2 µg/kg IV bolus at induction, followed by a continuous infusion of 1-2 µg/kg/h during maintenance of anesthesia. Standard anesthesia will be provided with propofol, rocuronium, and sevoflurane.
  Arms: Fentanyl Group
Drug: Remifentanil 1 µg/kg IV bolus + 0.1-1 µg/kg/min infusion during anesthesia — Patients will receive remifentanil 1 µg/kg IV bolus at induction, followed by a continuous infusion of 0.1-1 µg/kg/min during maintenance of anesthesia. Standard anesthesia will be provided with propofol, rocuronium, and sevoflurane.
  Arms: Remifentanil Group

SUMMARY:
Background: Postoperative ileus (POI) is a common complication after abdominal surgery, leading to delayed gastrointestinal recovery, prolonged hospitalization, and increased healthcare costs. Opioids, while essential for intraoperative analgesia, are known to impair bowel motility through their μ-receptor effects. Among opioids, fentanyl and remifentanil are widely used but differ in their pharmacokinetic and pharmacodynamic profiles. Remifentanil undergoes rapid metabolism, resulting in a shorter context-sensitive half-life, while fentanyl accumulates with longer infusions. Although remifentanil may theoretically have less impact on bowel recovery, its potential to induce opioid-induced hyperalgesia (OIH) and increased analgesic requirements might prolong gastrointestinal dysfunction and worsen postoperative pain outcomes.

Objective: This randomized controlled trial aims to compare the effects of intraoperative fentanyl versus remifentanil on the recovery of postoperative bowel function and pain outcomes in patients undergoing elective laparoscopic cholecystectomy.

Methods: A total of 106 patients, aged 18-65 years and classified as ASA I-II, will be randomized into two groups: Group F (fentanyl) and Group R (remifentanil). Standardized anesthesia with propofol, rocuronium, and sevoflurane will be applied. The primary endpoint is time to first flatus. Secondary endpoints include time to first defecation, tolerance of oral diet, incidence of prolonged POI, postoperative pain scores, analgesic consumption, PONV incidence, PACU and hospital length of stay, and patient satisfaction.

Significance: The findings of this study will provide clinical evidence on whether fentanyl or remifentanil is more advantageous in terms of gastrointestinal recovery and pain management following laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* American Society of Anesthesiologists (ASA) physical status I or II
* Scheduled for elective laparoscopic cholecystectomy
* Provided written informed consent

Exclusion Criteria:

* Opioid use preoperatively
* Previous abdominal surgery
* History of ileus or gastrointestinal disease
* Preoperative electrolyte imbalance
* Liver or renal failure
* Neuromuscular or psychiatric disorders
* Known allergy to study medications
* Emergency surgery
* Surgical duration exceeding 90 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to first flatus | Up to 72 hours postoperatively
  Time from admission to the post-anesthesia care unit (PACU) until the first passage of flatus, recorded in hours.

SECONDARY OUTCOMES:
Time to first defecation | Up to 72 hours postoperatively
  Time from postoperative care unit admission to first defecation, recorded in hours.
Postoperative pain scores (NRS) | First 24 hours postoperatively
  Pain intensity assessed using Numeric Rating Scale (0-10) at 0, 2, 4, 6, 12, and 24 hours after surgery.
Incidence of prolonged postoperative ileus | Within 7 days postoperatively
  Defined as persistence of ≥2 of the following for more than 3 days postoperatively: nausea/vomiting, absence of flatus for 24h, inability to tolerate oral diet for 24h, abdominal distension, radiological confirmation.
Rescue analgesic consumption | First 24 hours postoperatively
  Total amount of tramadol administered for NRS ≥4.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niedermayer S, Heyn J, Guenther F, Kuchenhoff H, Luchting B. Remifentanil for abdominal surgery is associated with unexpectedly unfavorable outcomes. Pain. 2020 Feb;161(2):266-273. doi: 10.1097/j.pain.0000000000001713. PMID 31592999
- [Background] de Boer HD, Detriche O, Forget P. Opioid-related side effects: Postoperative ileus, urinary retention, nausea and vomiting, and shivering. A review of the literature. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):499-504. doi: 10.1016/j.bpa.2017.07.002. Epub 2017 Jul 8. PMID 29739538
- [Background] Muller-Lissner S, Bassotti G, Coffin B, Drewes AM, Breivik H, Eisenberg E, Emmanuel A, Laroche F, Meissner W, Morlion B. Opioid-Induced Constipation and Bowel Dysfunction: A Clinical Guideline. Pain Med. 2017 Oct 1;18(10):1837-1863. doi: 10.1093/pm/pnw255. PMID 28034973
- [Background] Vather R, Trivedi S, Bissett I. Defining postoperative ileus: results of a systematic review and global survey. J Gastrointest Surg. 2013 May;17(5):962-72. doi: 10.1007/s11605-013-2148-y. Epub 2013 Feb 2. PMID 23377782